CLINICAL TRIAL: NCT00227370
Title: A Phase III, Randomized, Double-Blind Comparison of Oral Valganciclovir and Placebo for Prevention of CMV After Lung Transplantation
Brief Title: Comparison of Oral Valganciclovir and Placebo for the Prevention of Cytomegalovirus (CMV) After Lung Transplantation
Acronym: Valgan
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Pro00013245; 4623 (Val038) (Other: Alternative study ID)
Record Dates: First submitted 2005-09-26; First posted 2005-09-28 (Estimated); Results first posted 2013-04-29 (Estimated); Last update posted 2024-10-04 (Actual); Status verified 2024-09

CONDITIONS: Cytomegalovirus Infections
Keywords: Acute rejection; Non-CMV infections; Resistance
MeSH Terms: conditions — Cytomegalovirus Infections | interventions — Valganciclovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- 1 (Active Comparator): Valganciclovir 900 mg QD for 9 months post lung transplant.
  Interventions: Drug: valganciclovir
- 2 (Placebo Comparator): placebo for 9 months post lung transplant
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: valganciclovir — valgan 900mg QD x 9 months post lung transplant
  Other Names: valcyte
  Arms: 1
Other: Placebo
  Arms: 2

SUMMARY:
The study evaluated the efficacy and safety of a prolonged, continuous course of Valganciclovir (Valgan) in the prevention of CMV by comparing 3 months of Vaglanciclovir, the standard of care upon initiation of the study, to 12 months of Valganciclovir.

DETAILED DESCRIPTION:
A multi-center two phase, double-blind, placebo controlled, randomized prospective study of 130 lung transplant recipients. Patients will be screened and consented prior to transplant. All consented patients will receive IV ganciclovir within 24 hours of transplant for not more than 14 days. Patients will enroll in Phase I of the study is an open label safety and efficacy analysis of three months of oral valganciclovir in adult transplant recipients who are at risk for CMV. After completion of 3 months of open label therapy, patients that meet the criteria for Phase II of the study will be randomized to 9 months of blinded therapy (Placebo/Valgan). Phase II of the study is designed to assess the efficacy of short course sequential IV ganciclovir followed by oral valganciclovir as compared to the extended period of oral valganciclovir prophylaxis in the prevention of CMV disease in at risk lung transplant recipients

ELIGIBILITY:
Inclusion Criteria for Phase I:

* Adult lung transplant recipients age 18 or older
* At risk for CMV (donor or recipient serology must be positive for CMV)
* Adequate hematological and renal function,
* On intravenous (IV) ganciclovir within 24 hours of surgery
* Agreement to use effective methods of contraception
* Negative pregnancy
* Tolerate oral medications within 2 weeks of transplant
* Negative baseline CMV PCR
* Able to understand and sign the informed consent

Exclusion Criteria for Phase 1:

* Repeat transplantation
* Mechanical ventilation at study entry
* Oral or intravenous ganciclovir treatment outside the study protocol
* Invasive fungal infection
* Participation in another investigational study
* Acute CMV infection or disease
* Anti-CMV therapy within 30 days before enrollment
* Uncontrolled diarrhea or malabsorption
* Allergic reaction to study drug
* Required use of prohibited medications
* Lactating women
* Pregnancy
* Renal failure

Inclusion Criteria for Phase II:

* Negative serial post transplant PCRs at day 75
* Negative bronchial cultures for CMV
* Adequate hematological and renal function at day 75
* IV ganciclovir for up to 2 weeks post operation and open label up to day 90
* Effective contraceptives
* Negative pregnancy

Exclusion Criteria Phase II:

* Renal failure
* Serious adverse events (SAE) related to study drug
* CMV disease (study endpoint)
* Withdraw consent for Phase II

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2003-07; Primary Completion 2008-04 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott M Palmer, MD, Principal Investigator — Duke University
Locations (1):
- DukeUMC, Durham, North Carolina, United States

REFERENCES:
- [Derived] Vernooij RW, Michael M, Colombijn JM, Owers DS, Webster AC, Strippoli GF, Hodson EM. Pre-emptive treatment for cytomegalovirus viraemia to prevent cytomegalovirus disease in solid organ transplant recipients. Cochrane Database Syst Rev. 2025 Jan 14;1(1):CD005133. doi: 10.1002/14651858.CD005133.pub4. PMID 39807668
- [Derived] Vernooij RW, Michael M, Ladhani M, Webster AC, Strippoli GF, Craig JC, Hodson EM. Antiviral medications for preventing cytomegalovirus disease in solid organ transplant recipients. Cochrane Database Syst Rev. 2024 May 3;5(5):CD003774. doi: 10.1002/14651858.CD003774.pub5. PMID 38700045
- [Derived] Palmer SM, Limaye AP, Banks M, Gallup D, Chapman J, Lawrence EC, Dunitz J, Milstone A, Reynolds J, Yung GL, Chan KM, Aris R, Garrity E, Valentine V, McCall J, Chow SC, Davis RD, Avery R. Extended valganciclovir prophylaxis to prevent cytomegalovirus after lung transplantation: a randomized, controlled trial. Ann Intern Med. 2010 Jun 15;152(12):761-9. doi: 10.7326/0003-4819-152-12-201006150-00003. PMID 20547904

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Prospective subjects were screened and enrolled from July 2003 - January 2007 at 11 US lung transplant centers. 189 subjects were screened and 157 met inclusion criteria and were therefore enrolled in the study.
Pre-assignment Details: Upon receipt of a lung transplant, enrolled subjects received 90 days of valganciclovir for CMV prophylaxis, per standard of care, and then were randomly assigned, 1:1, in a double blind fashion, to either the extended prophylaxis group (9 additional months of standard of care dosing Valganciclovir, adjusted for renal function) or placebo group.
Groups:
- Placebo Group: Upon randomization at 3 months, patients discontinued Valganciclovir and received no CMV prophylaxis for the next 9 months (short course prophylaxis). 3 months of Valganciclovir was the standard of care for CMV prevention at the time of study initiation. This was the prespecified placebo group/intervention arm.
- Treatment Group: Upon randomization at 3 months, patients remained on Valganciclovir for 9 additional months (extended course prophylaxis).
Period: Overall Study
Arm/Group | Placebo Group | Treatment Group
Started | 66 (Placebo Group) | 70 (Treatment Group)
Completed | 45 | 46
Not Completed | 21 | 24
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Death | 3 | 4
Not completed — Adverse Event | 6 | 11
Not completed — Physician Decision | 9 | 6
Not completed — Other reasons | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo Group: Upon randomisation at 3 months, patients discontinued Valganciclovir and received no CMV prophylaxis
- Treatment Group: Upon randomisation at 3 months, patients remained on Valganciclovir for 9 additional months.
- Total: Total of all reporting groups
Arm/Group | Placebo Group | Treatment Group | Total
Number analyzed (Participants) | 66 | 70 | 136
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age | 50.6 (13.8) | 51.9 (12.2) | 51.3 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 41 | 69
  Male | 38 | 29 | 67
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 7 | 13
  White | 60 | 63 | 123
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
FEV1, liters [Median (Inter-Quartile Range); unit: liters] — Forced Expiratory Volume in 1 second, liters
  liters | 0.75 [0.53 to 1.32] | 0.80 [0.64 to 1.23] | 0.79 [0.57 to 1.24]
Indication for Lung Transplant [Number; unit: subjects] — Placebo Group: Treatment Group:
  COPD: 35 33 Cystic Fibrosis: 11 12 IPF: 16 16 Sarcoid: 2 3 Other: 2 6
  subjects
    COPD | 35 | 33 | 68
    Idiopathic Pulmonary Fibrosis | 16 | 16 | 32
    Cystic Fibrosis | 11 | 12 | 23
    Sarcoid | 2 | 3 | 5
    Other | 2 | 6 | 8
FVC, liters [Median (Inter-Quartile Range); unit: liters] — forced vital capacity
  liters | 2.02 [1.52 to 2.62] | 1.89 [1.49 to 2.32] | 1.95 [1.51 to 2.48]
6MWD, feet [Median (Inter-Quartile Range); unit: feet] — the distance in feet a subject walks in 6 minutes
  feet | 1168 [946 to 1350] | 1120 [945 to 1380] | 1155 [945 to 1380]
Smoking History [Number; unit: subjects] — Placebo Treatment Past:44/66 49/70 Current: 0 0 No hx:22/66 21/70
  subjects
    No Smoking History/Never Smoked (past or present) | 22 | 21 | 43
    Past Smoking History: former smokers who quit | 44 | 49 | 93
    Current Smoking | 0 | 0 | 0
Daily Supplemental Oxygen Use [Number; unit: subjects] — the number of subjects requiring supplemental daily oxygen through nasal canula or face mask.
  subjects
    Supplemental Oxygen use | 53 | 51 | 104
    No supplemental oxygen use | 13 | 19 | 32

OUTCOME MEASURES:

1. Primary Outcome: Incidence of CMV End Organ Disease
Description: The primary study end point was CMV end-organ disease determined by positive tissue immunostain or characteristic histopathology assessed for within 300 days post randomization.
Time Frame: over the course of 300 days after randomization
Population: Intention to treat analysis was conducted.
Measure: Number; unit: participants
Groups:
- Placebo Group: Upon randomization at 3 months, patients discontinued Valganciclovir and received no CMV prophylaxis for the next 9 months (short course prophylaxis)
Arm/Group | Placebo Group | Treatment Group
Number analyzed (Participants) | 66 | 70
participants | 21 | 1

2. Primary Outcome: Incidence of CMV Syndrome
Description: CMV clinical syndrome, with either positive serum PCR or positive culture for CMV from bronchoalveolar lavage and at least 2 of the following: fever, leukopenia, thrombocytopenia, elevated liver function test results malaise, reduction in pulmonary function (FEV1) greater than 20percent of baseline, or radiographic infiltrate consistent with CMV (all in the absence of other causes)
Time Frame: over the course of 300 days after randomization
Population: intention to treat analysis
Measure: Number; unit: participants
Arm/Group | Placebo Group | Treatment Group
Number analyzed (Participants) | 66 | 70
participants | 13 | 0

3. Secondary Outcome: Any CMV Infection
Description: Inclusive of CMV syndrome, disease, or infection not meeting primary end point.
Time Frame: over the course of 300 days post randomization
Population: intention to treat
Measure: Number; unit: participants
Arm/Group | Placebo Group | Treatment Group
Number analyzed (Participants) | 66 | 70
participants | 42 | 7

4. Secondary Outcome: Biopsy Proven Acute Lung Rejection
Time Frame: over the course of 300 days of randomization
Population: intention to treat
Measure: Number; unit: participants
Arm/Group | Placebo Group | Treatment Group
Number analyzed (Participants) | 66 | 70
participants | 22 | 15

5. Secondary Outcome: Non-CMV Infection
Description: non cmv opportunistic infections
Time Frame: over the course of 300 days after randomization
Population: intention to treat
Measure: Number; unit: participants
Arm/Group | Placebo Group | Treatment Group
Number analyzed (Participants) | 66 | 70
participants | 35 | 38

6. Secondary Outcome: Severity of Viremia
Description: upon diagnosis of cmv disease, the number of CMV DNA copies/mL as measured by PCR
Time Frame: over the course of 300 days after randomization
Population: Intention to treat
Measure: Median (Inter-Quartile Range); unit: CMV copies/mL
Arm/Group | Placebo Group | Treatment Group
Number analyzed (Participants) | 66 | 70
CMV copies/mL | 110,000 [40,000 to 361,569] | 3,200 [2,700 to 3,700]

7. Secondary Outcome: Ganciclovir Resistance
Description: UL97 genotyping was done on all positive samples for CMV DNA at 1000 copies/mL, with resistance defined by the presence of 1 or more mutations shown by marker transfer to confer phenotypic ganciclovir resistance
Time Frame: over the course of 300 days post randomization
Population: intention to treat
Measure: Number; unit: participants
Arm/Group | Placebo Group | Treatment Group
Number analyzed (Participants) | 66 | 70
participants | 1 | 2

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the first day posttransplant to the close of the study (day 390); however they were stratified by Phases (I and II) therefore SAEs are only reported for phase II subjects (ie only randomized subjects).
Arm/Group | Placebo Group | Treatment Group
Serious Adverse Events (participants affected / at risk) | 35/66 | 38/70
Other Adverse Events (participants affected / at risk) | 64/66 | 70/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Group (N=66) | Treatment Group (N=70)
SEPSIS (Infections and infestations) | 0 | 1
GASTROENTERITIS (Gastrointestinal disorders) | 0 | 3
CLOSTRIDIUM DIFFICILE COLITIS (Gastrointestinal disorders) | 1 | 0
CYTOMEGALOVIRUS COLITIS (Infections and infestations) | 1 | 0
WOUND INFECTION (Infections and infestations) | 1 | 0
PLEURAL EFFUSION (Infections and infestations) | 2 | 0
RESPIRATORY FAILURE (Infections and infestations) | 1 | 1
ACUTE RESPIRATORY DISTRESS SYNDROME (General disorders) | 0 | 1
BRONCHOSTENOSIS (General disorders) | 0 | 1
LUNG INFILTRATION (Infections and infestations) | 0 | 1
PULMONARY HAEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 0 | 1
LUNG TRANSPLANT REJECTION (Immune system disorders) | 5 | 4
TRANSPLANT REJECTION (Immune system disorders) | 3 | 2
GASTROINTESTINAL DISORDERS (Gastrointestinal disorders) | 7 | 3
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 1
VOMITING (Gastrointestinal disorders) | 1 | 1
GASTROINTESTINAL DISORDER (Gastrointestinal disorders) | 1 | 0
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 | 0
NEUTROPENIA (Immune system disorders) | 3 | 9
ANAEMIA (Blood and lymphatic system disorders) | 1 | 2
PYREXIA (Gastrointestinal disorders) | 1 | 3
MULTI-ORGAN FAILURE (General disorders) | 0 | 1
CARDIAC DISORDERS (Cardiac disorders) | 2 | 5
CARDIAC ARREST (Cardiac disorders) | 1 | 0
ENCEPHALOPATHY (Vascular disorders) | 0 | 2
HEADACHE (General disorders) | 0 | 1
ISCHAEMIC STROKE (Blood and lymphatic system disorders) | 0 | 1
Opportunistic Infections, all organ systems (Infections and infestations) | 31 | 32
Opportunistic Infections, all organ systems, mild (Infections and infestations) | 11 | 8
Opportunistic Infections, all organ systems, moderate (Infections and infestations) | 17 | 17
Opportunistic Infections, all organ systems, severe (Infections and infestations) | 3 | 7
Hospitalization (Cardiac disorders) | 0 | 1
Death (Infections and infestations) | 3 | 4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Group (N=66) | Treatment Group (N=70)
RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS (Respiratory, thoracic and mediastinal disorders) | 38 | 42
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 10 | 16
cough (Respiratory, thoracic and mediastinal disorders) | 14 | 8
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 7 | 11
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 7 | 11
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 6 | 6
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 5 | 5
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 3 | 7
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 4 | 4
LUNG INFILTRATION (Respiratory, thoracic and mediastinal disorders) | 2 | 4
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 2 | 4
BRONCHOSTENOSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 5
OEDEMA PERIPHERAL (Respiratory, thoracic and mediastinal disorders) | 12 | 17
FATIGUE (Respiratory, thoracic and mediastinal disorders) | 13 | 15
PYREXIA (Respiratory, thoracic and mediastinal disorders) | 11 | 7
CHEST PAIN (Respiratory, thoracic and mediastinal disorders) | 8 | 6
CHEST DISCOMFORT (Respiratory, thoracic and mediastinal disorders) | 3 | 6
MALAISE (Respiratory, thoracic and mediastinal disorders) | 4 | 3
OEDEMA (Respiratory, thoracic and mediastinal disorders) | 4 | 3
CHILLS (Respiratory, thoracic and mediastinal disorders) | 4 | 2
ASTHENIA (Respiratory, thoracic and mediastinal disorders) | 0 | 4
GENERALISED OEDEMA (Respiratory, thoracic and mediastinal disorders) | 3 | 0
GASTROINTESTINAL DISORDERS (Gastrointestinal disorders) | 35 | 41
DIARRHOEA (Gastrointestinal disorders) | 13 | 14
VOMITING (Gastrointestinal disorders) | 9 | 11
NAUSEA (Gastrointestinal disorders) | 7 | 11
ABDOMINAL PAIN (Gastrointestinal disorders) | 4 | 8
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 4 | 8
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 5 | 5
CONSTIPATION (Gastrointestinal disorders) | 6 | 4
UPPER RESPIRATORY TRACT INFECTION (Respiratory, thoracic and mediastinal disorders) | 12 | 10
PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 9 | 4
SINUSITIS (Respiratory, thoracic and mediastinal disorders) | 6 | 6
BRONCHITIS (Respiratory, thoracic and mediastinal disorders) | 2 | 4
SEPSIS (Respiratory, thoracic and mediastinal disorders) | 1 | 4
HEADACHE (Nervous system disorders) | 12 | 11
TREMOR (Nervous system disorders) | 7 | 4
DIZZINESS (Nervous system disorders) | 4 | 5
HYPOAESTHESIA (Nervous system disorders) | 2 | 4
MIGRAINE (Nervous system disorders) | 4 | 0
SINUS HEADACHE (Nervous system disorders) | 4 | 0
WEIGHT INCREASED (Investigations) | 6 | 6
PULMONARY FUNCTION TEST DECREASED (Investigations) | 2 | 4
HEPATIC ENZYME INCREASED (Investigations) | 1 | 4
BREATH SOUNDS ABNORMAL (Investigations) | 0 | 4
ANAEMIA (Blood and lymphatic system disorders) | 5 | 15
LEUKOPENIA (Blood and lymphatic system disorders) | 5 | 14
NEUTROPENIA (Blood and lymphatic system disorders) | 3 | 9
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 | 4
LUNG TRANSPLANT REJECTION (Immune system disorders) | 18 | 18
TRANSPLANT REJECTION (Immune system disorders) | 5 | 4
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 7 | 6
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 10 | 3
BACK PAIN (Musculoskeletal and connective tissue disorders) | 5 | 4
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 2 | 6
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 5 | 3
HYPERKALAEMIA (Metabolism and nutrition disorders) | 6 | 1
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 2 | 4
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 | 4
DEHYDRATION (Metabolism and nutrition disorders) | 4 | 1
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 4 | 1
ALOPECIA (Skin and subcutaneous tissue disorders) | 6 | 4
rash (Skin and subcutaneous tissue disorders) | 6 | 0
HYPERTENSION (Vascular disorders) | 7 | 11
RENAL FAILURE (Renal and urinary disorders) | 0 | 10
RENAL FAILURE ACUTE (Renal and urinary disorders) | 3 | 5
INSOMNIA (Psychiatric disorders) | 7 | 4
DEPRESSION (Psychiatric disorders) | 4 | 4
VISION BLURRED (Eye disorders) | 3 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No